CLINICAL TRIAL: NCT02377557
Title: Topical Steroid Registry: Observational Study to Assess Safety and Use Pattern in Korea
Brief Title: Observational Study to Assess Safety and Utility Pattern of Topical Steroids
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Collaborators: Korean Ministry of Food and Drug Safety (Unknown); College of Pharmacy, Seoul National University (Unknown)
Responsible Party: Principal Investigator, Ju-Yeun Lee, Ph.D, Hanyang University
Other Study IDs: MFDS2014-20384
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Skin Diseases
Keywords: Dermatologic Agent
MeSH Terms: conditions — Skin Diseases | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topical Steroids

SUMMARY:
To assess incidence of adverse drug reactions and use pattern of topical steroids among patients who are prescribed or purchase over the counter (OTC) topical steroids for skin conditions in Korea

DETAILED DESCRIPTION:
* Active collection of safety data, systemic and local adverse events.
* In addition to spontaneous adverse event reports, patients will be asked on occurrence of adverse events upon use of topical steroids at 1 month, 2 month, and 6 month after study enrollment by e-mail or phone call
* Causality of adverse events will be assessed by independent two professionals
* Document the utility pattern of topical steroid, misuse (inappropriate indication) or overuse (in terms of application frequency or treatment duration)
* Collection of information related with adverse event management

ELIGIBILITY:
Inclusion Criteria:

* All patients or guardian of child purchased topical steroids in Korea
* Informed consent to participate
* Willing to follow and abide by the protocol

Exclusion Criteria:

* None

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients or guardian of child purchased topical steroids in Korea
Sampling Method: Non-Probability Sample
Enrollment: 1175 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of adverse drug reaction upon use of topical steroid | 4 week after time of enrollment

SECONDARY OUTCOMES:
Rate of adverse drug reaction upon use of topical steroid | 2 month after time of enrollment
Rate of adverse drug reaction upon use of topical steroid | 6 month after time of enrollment
Rate of adverse drug reaction by potency, route of purchase (prescription/self diagnosed), drug classification (prescription only/over the counter) | 1 month after time of enrollment
Rate of misuse and overuse of topical steroids | 6 month after time of enrollment
Impact of covariates on incidence of adverse drug reaction | 6 month after time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Yeun Lee, Ph.D., Principal Investigator — College of Pharmacy, Hanyang University
Locations (1):
- College of Pharmacy, Hanyang University, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No